CLINICAL TRIAL: NCT06667674
Title: Efficacy and Mechanisms of Change of Online Cognitive Behavioural Therapy for Prolonged Grief Disorder After Loss: a Three-armed Randomised Control Trial
Brief Title: A Swedish Internet CBT for Prolonged Grief Disorder: a Three-armed RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-02632-01
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Prolonged Grief Disorder
MeSH Terms: conditions — Prolonged Grief Disorder

STUDY DESIGN:
Intervention Model Description: Active control group, waitlist control group and intervention group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention group (Experimental): Participants will receive cognitive behavioral therapy treatment (iCBT) for prolonged grief.
  Interventions: Behavioral: iCBT for prolonged grief
- Active control (Active Comparator): Participants will receive psychoeducation about grief and common grief reactions.
  Interventions: Behavioral: Active control
- Waitlist control (No Intervention): Participants will be offered the iCBT treatment for prolonged grief after 10 weeks.

INTERVENTIONS:
Behavioral: iCBT for prolonged grief — Participants will undergo a 10-week internet-delivered, therapist-led cognitive behavioral therapy treatment (iCBT) for prolonged grief, which includes psychoeducation about grief and common grief reactions, exposure, cognitive restructuring and behavioral activation.
  Arms: Intervention group
Behavioral: Active control — Participants will undergo a 10-week internet-delivered, therapist-led treatment, which includes psychoeducation about grief and common grief reactions.
  Arms: Active control

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of internet-delivered Cognitive Behavioral Therapy (iCBT) in reducing symptoms of prolonged grief in adults diagnosed with prolonged grief disorder.

The main questions the study aims to answer are:

* Does iCBT reduce symptoms of prolonged grief disorder, posttraumatic stress, and depression following the death of a loved one in the short and long term?
* What mechanisms contribute to the effectiveness of iCBT in treating prolonged grief disorder?

The iCBT intervention will be compared to a waitlist control group and an active control group to see if iCBT reduces symptoms of prolonged grief disorder more effectively than no treatment or a placebo treatment.

Participants will:

* Be randomly assigned to either the iCBT group, an active control group or a waitlist control group
* Complete online assessments of symptom severity, grief cognitions, and level of avoidance before, during and after intervention
* Engage in 10 weeks of a therapist-guided online treatment

DETAILED DESCRIPTION:
The death of a loved one can lead to various mental and physical health problems. Previous research has shown that Cognitive Behavioral Therapy (CBT) can be effective in recuding symptoms of prolonged grief. However, most previous studies have had small sample sizes and lacked follow-up assessments over time.

The purpose of this project is to conduct a large randomized controlled trial (RCT) to evaluate the effectiveness of internet-delivered cognitive-behavioral therapy (iCBT) in reducing symptoms of prolonged grief, depression, and posttraumatic stress in adults who have lost a loved one. The iCBT treatment will be compared against both an active control condition and a waitlist condition. Participants in the active control condition will receive a simplified version of the iCBT treatment, which is also therapist-led but lacks active CBT components. The waitlist control group will receive the iCBT treatment after 10 weeks. Follow-up assessments will be conducted at 6 and 12 months after treatment completion.

The study will also examine potential moderators (such as baseline symptom levels and loss characteristics) and mediators (such as belief in treatment efficacy, changes in negative cognitions and level of avoidance) on treatment effects. This may provide insights into the effectiveness of prolonged grief treatment and factors that influence treatment outcomes.

Participants will be recruited through advertisements on social media platforms, and organisations and clinical contacts. Individuals interested in participating in the study register their interest on a website linked to the research project, and complete an initial screening form. Potential participants are contacted by phone to schedule an assessment interview over video, which includes the structured diagnostic interview Mini International Neuropsychiatric Interview (M.I.N.I.). Subsequently, eligible participants are randomized to iCBT, active control, or waitlist control. The participants will be informed that they have been randomly assigned to either a waitlist or one of two grief treatment programs but will not know which of the treatments they are in, and are thus blind at the beginning of the study. The treatment is accessed on a digital platfom.

This study is the first of its kind in Sweden to examine the effectiveness of internet-delivered treatment for prolonged grief. Additionally, it is the first trial to assess both short- and long-term effects of iCBT for prolonged grief compared to an active control group.

ELIGIBILITY:
Inclusion Criteria:

* Currently residing in Sweden
* Lost a relative or close friend to any cause of death at least six months ago
* Suffers from prolonged grief disorder

Exclusion Criteria:

* Ongoing severe psychiatric problems that may prevent treatment implementation or require more urgent care (e.g., participants with untreated psychotic disorder, untreated bipolar disorder, ongoing substance abuse, elevated suicide risk)
* Change in dosage of any medication for mental health issues (e.g., antidepressant medication) in the past four weeks or in the next two months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change (from baseline) in Traumatic Grief Inventory Self Report Plus, TGI-SR+ | 0, 5 and 10 weeks. Follow-up at 6 and 12 months post-treatment.
  A 22-item, self-rated measure of prolonged grief symptoms. Total score ranges from 22 to 110, where a higher score indicates more symptoms.

SECONDARY OUTCOMES:
Change (from baseline) in Posttraumatic stress disorder checklist for DSM-5, PCL-5 | 0, 5 and 10 weeks. Follow-up at 6 and 12 months post-treatment.
  A 20-item, self-rated measure of posttraumatic stress disorder. Total score ranges from 0-80, and a higher score indicates more symptoms
Change (from baseline) in Patient Health Questionnaire, PHQ-9 | 0, 5 and 10 weeks. Follow-up at 6 and 12 months post-treatment.
  A 9-item, self-rated measure of depression. Total score ranges from 0-27, and a higher score indicates more symptoms
Change (from baseline) in Depressive and Anxious Avoidance in Prolonged Grief questionnaire, DAAPGQ | 0, 5 and 10 weeks. Follow-up at 6 and 12 months post-treatment.
  A 9-item, self-rated measure of avoidance. Total score ranges from 9-72, and a higher score indicates more avoidance
Change (from baseline) in Grief Cognitions Questionniare, GCQ | 0, 5 and 10 weeks. Follow-up at 6 and 12 months post-treatment.
  An 18-item, self-rated measure of grief cognitions. Total score ranges from 0-90, and a higher score indicates more grief cognitions
Change (from baseline) in the short version of Traumatic Grief Inventory Self Report Plus, Short version TGI-SR+ | Weekly assessments between week 0 and week 10, excluding week 5.
  Five items from TGI-SR+, measuring PGD symptoms. Total score ranges from 5-25, and a higher score indicates more symptoms.
Change (from baseline) in Short Form Posttraumatic stress disorder checklist for DSM-5, Short form PCL-5 | Weekly assessments between week 0 and week 10, excluding week 5.
  Four items from PCL-5, measuring PTSD symptoms. Total score ranges from 0-16, and a higher score indicates more symptoms.
Change (from baseline) in Patient Health Questionnaire, PHQ-2 | Weekly assessments between week 0 and week 10, excluding week 5.
  Two items from PHQ-9, measuring depression. Total score ranges from 0-6, and a higher score indicates more symptoms.

OTHER OUTCOMES:
Demographics | 0 months
  Age, gender, time since loss, marital status, employment status, loss-related variables
Treatment Credibility Scale, TCS | Week 2
  A 5-item, self-rated measure of participants' view of treatment credibility. Total score ranges from 5-50, and higher scores indicate stronger beliefs in treatment efficacy and credibility.
Negative effects questionnaire | Week 10
  Negative effects questionnaire (NEQ; Rozental et al., 2019)
Client Satisfaction Questionnaire Eight, CSQ-8 | Week 10
  An 8-item, self-rated measure of participants' treatment experience. Total score ranges from 8-32, where a higher score indicates greater satisfaction with the treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Region Uppsala, KBT via nätet, Nära vård digitalt, Uppsala
  - Uppsala university, Dep of Womens and Childrens Health, Uppsala